CLINICAL TRIAL: NCT01754376
Title: COMBAT 1: A Phase II Trial of Combined BRAF-Targeted Therapy and Immunotherapy for Melanoma
Brief Title: Combined BRAF-Targeted Therapy & Immunotherapy for Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: changes in available treatments for melanoma
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ryan Sullivan, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-343
Record Dates: First submitted 2012-12-16; First posted 2012-12-21 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-01

CONDITIONS: Melanoma
Keywords: Metastatic; Unresectable; V600E mutation
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — aldesleukin; Interleukin-2; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Oral vemurafenib 960 milligrams twice a day plus intravenous aldesleukin 600,000 IU/kg every eight hours to tolerance (maximum 14 doses) over five days on days 15-19 of cycle 1 and on days 1-5 of cycle 2. (A cycle is 28 days)
  The first course of treatment will consist of three 28-day cycles (12 weeks): 2 weeks of lead-in vemurafenib plus 3 weeks on IL-2 plus 7 weeks wait.
  A second course may be given at the discretion of the investigator, if there is evidence of tumor stability or regression.
  Interventions: Drug: Aldesleukin; Drug: Vemurafenib

INTERVENTIONS:
Drug: Aldesleukin — Intravenous therapy given every 8 hours for up to 14 doses per week.
  Other Names: Interleukin 2; IL-2; Proleukin
Drug: Vemurafenib — Tablets given twice daily.
  Other Names: Zelboraf; PLX4032; RG7204; RO5185426

SUMMARY:
This research study is a Phase II clinical trial of an investigational combination of drugs (vemurafenib and aldesleukin) to learn whether the combination works in treating a specific cancer. While both vemurafenib and aldesleukin are approved by the FDA for the treatment of metastatic melanoma, the FDA has not yet approved the combination of vemurafenib and aldesleukin.

Researchers have found that a large number of melanoma cells have mutations in the BRAF gene. It has been shown that vemurafenib blocks the effects of these mutations in the BRAF gene, and, as a result, may help to prevent cancer growth.

Aldesleukin, also referred to as IL-2, is an immunotherapy drug administered via IV infusion that increases the growth of key cells within the immune system that are responsible for targeting cancer cells. Activating more of these key cells, called T-lymphocytes and natural-killer cells, leads to increased cancer cell death.

The BRAF gene is located on a larger pathway called the MAPK pathway. Studies have shown that when a BRAF inhibitor, like vemurafenib is used to block the MAPK pathway, melanocytes, or cancer cells express more proteins on their surfaces, making them easier for T-lymphocytes and natural killer cells to recognize and kill them. This suggests that combining BRAF-targeted therapy with aldesleukin, which activates more of these white blood cells, can lead to an increase in the death of cancer cells.

In this research study, the investigators are looking to see whether the combination of vemurafenib (a BRAF-inhibitor) combined with aldesleukin(an immunotherapy drug) work together to produce a better health outcome in people with metastatic melanoma.

DETAILED DESCRIPTION:
Subjects will take oral vemurafenib twice a day for 2 weeks. Following this lead-in period, subjects will receive aldesleukin via IV infusion on Day 15 of the study. One course of aldesleukin is 12 weeks long; subjects will receive aldesleukin via IV infusion every 8 hours for the first five days. Subjects will be hospitalized for the 5 days that they are receiving aldesleukin.

Week 1 of aldesleukin will be days 15-19 (M-F) of the 12 week cycle. Following Week 1 of therapy, subjects will be discharged from the hospital and only take vemurafenib at home for the following week. Subjects will then come in for one more week of aldesleukin during days 29-33 of the 12 week cycle. This is referred to as Week 2 of aldesleukin.

Subjects will continue to take vemurafenib twice daily during the course of aldesleukin. Their cancer will be evaluated at screening and at Week 12 following the beginning of the first aldesleukin course with a CT scan. After the first cycle, tumors will be evaluated every 8 weeks for the first year, then every 12 weeks for years 2 and 3, every 6 months for year 5, and annually thereafter.

If scans show that the subject's cancer has improved after the first course of aldesleukin, subjects may be allowed to continue on to a second course. In the event of a second course of aldesleukin, subjects will remain on vemurafenib throughout the second course.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or unresectable melanoma with V600E mutation
* Measurable disease
* May have received prior immunotherapy (excluding interleukin 2)
* Life expectancy greater than 3 months
* Recovered from effects of previous surgery and/or traumatic injury
* Must agree to use effective contraception

Exclusion Criteria:

* Pregnant or breastfeeding
* Psychological, familial or other conditions that could hamper compliance with protocol
* Receiving other study agents
* History of carcinomatous meningitis
* Known active brain metastases
* Have received a BRAF inhibitor
* Uncontrolled intercurrent illness
* HIV positive on antiretroviral therapy
* History of a different malignancy within past 5 years (except cervical cancer in situ or basal/squamous cell carcinoma of the skin)
* Active hepatitis B or C
* Have received allogenic bone marrow transplant or organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-01; Primary Completion 2015-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Sullivan, MD, Principal Investigator — MGH Cancer Center
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
All raw analytic data on tumor and blood samples will be shared, upon acceptance of manuscript.

REFERENCES:
- [Derived] Mooradian MJ, Reuben A, Prieto PA, Hazar-Rethinam M, Frederick DT, Nadres B, Piris A, Juneja V, Cooper ZA, Sharpe AH, Corcoran RB, Flaherty KT, Lawrence DP, Wargo JA, Sullivan RJ. A phase II study of combined therapy with a BRAF inhibitor (vemurafenib) and interleukin-2 (aldesleukin) in patients with metastatic melanoma. Oncoimmunology. 2018 Feb 1;7(5):e1423172. doi: 10.1080/2162402X.2017.1423172. eCollection 2018. PMID 29721378

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at Massachusetts General Hospital (Boston, MA) between February and November 2013
Groups:
- Treatment Arm: Oral vemurafenib twice a day IV infusion of aldesleukin
  Aldesleukin: Intravenous therapy given every 8 hours for up to 14 doses per week.
  Vemurafenib: Tablets given twice daily.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 6
Completed 2-week Lead in of Vemurafenib | 6
Completed | 3
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 42 [23 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Brain Metastasis present [Count of Participants; unit: Participants] | 1
ECOG Status [Count of Participants; unit: Participants] — The ECOG Scale of Performance Status describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability. A score of 0 indicates fully active, and a score of 5 indicates dead. (A score of one = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work)
  Participants
    ECOG Status = 0 | 3
    ECOG Status = 1 | 3
Previous treatments [Count of Participants; unit: Participants]
  Surgery | 6
  Adjuvant interferon-alfa | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: To assess the efficacy (as measured by progression-free survival (PFS)) of patients with metastatic melanoma with V600E mutation treated with the combination of vemurafenib and aldesleukin. Progression free survival is defined as the time between the first dose of study drug and the first occurrence of progression of disease or death from any cause. Progression is defined using Response Evaluation Criteria in Solid Tumors (RECIST v.1.1), as at least a 20% increase in the sum of the diameters of target lesions or the appearance of one or more new lesions.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
weeks | 35.8 [16 to 57]

2. Secondary Outcome: Overall Response Rate
Description: To determine the overall response rate (as defined as the rate of objective response (Complete Response (CR) or Partial Response (PR)) lasting continuously for 12 or more months, and beginning at any point within 12 months of initiating therapy) in patients treated with aldesleukin and vemurafenib. In this limited cohort, response rate was calculated as the proportion of patients with partial (PR) or complete response (CR) divided by the total number of patients treated. Per Response Evaluation Criteria in Solid Tumors (RECIST v.1.1), 'Complete Response' is the disappearance of all target lesions and 'Partial Response' is at least a 30% decrease in the sum of the diameters of target lesions, as measured via CT (computed tomography). Overally Response (OR) = CR + PR.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment Arm: Oral vemurafenib 960 milligrams twice a day plus intravenous aldesleukin 600,000 IU/kg every eight hours to tolerance (maximum 14 doses) over five days on days 15-19 of cycle 1 and on days 1-5 of cycle 2. (A cycle is 28 days)
  The first course of treatment will consist of three 28-day cycles (12 weeks): 2 weeks of lead-in vemurafenib plus 3 weeks on IL-2 plus 7 weeks wait.
  A second course may be given at the discretion of the investigator, if there is evidence of tumor stability or regression.
  Aldesleukin: Intravenous therapy given every 8 hours for up to 14 doses per week.
  Vemurafenib: Tablets given twice daily.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
percentage of participants | 83.3 [36 to 99]

3. Secondary Outcome: Overall Survival
Description: To determine the overall survival in patients treated with aldesleukin and vemurafenib. Overall survival is defined as the time between the first administration of study drug and death due to any cause.
Time Frame: 2 years
Population: Median overall survival was not reached
Measure: Median (Full Range); unit: months
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
months | NA [NA to NA] — Median overall survival was not reached

4. Secondary Outcome: Number of Participants Experiencing Grade 3 (Severe) Adverse Events
Description: To determine the toxicity and safety of concurrent administration of aldesleukin and vemurafenib by assessing adverse events experienced by participants.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
Participants | 6

5. Secondary Outcome: Mean Percentage of Aldesleukin Doses Received Per Participant
Description: To assess whether the number of doses of aldesleukin that can be safely administered is affected by the co-administration of vemurafenib. The total number of planned doses of aldesleukin was 28 in each of course 1 and course 2. A participant receiving all 28 doses in course 1 would be considered as receiving 100 percent of doses.
Time Frame: Approximately 9 months from start of treatment
Population: Six participants started course 1. Only 4 participants started course 2.
Measure: Mean (Full Range); unit: percentage of doses
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
percentage of doses
  Course 1 doses | 73 [61 to 86]
  Course 2 doses: number analyzed (Participants) | 4
  Course 2 doses | 54 [39 to 64]
  Total doses | 55 [32 to 70]

6. Secondary Outcome: Ratio of CD8+ T Cells to Regulatory T Cells
Description: Tumor samples were collected pre-treatment, after 1-2 weeks on vemurafenib alone and after administration of aldesleukin (high-dose interleukin 2, HD-IL2). Multi-parameter flow cytometry was performed to measure the frequency of regulatory T cells and of CD8+ T cells. The CD8/Treg ratio was calculated.
Time Frame: Up to 8 weeks from start of treatment
Population: Tumor tissue was only analyzed from one participant
Measure: Number; unit: ratio CD8/T reg cells
Arm/Group | Treatment Arm
Number analyzed (Participants) | 1
ratio CD8/T reg cells
  Pre-treatment | 43.9
  After vemurafenib alone | 20.5
  After aldesleukin | 4.04

ADVERSE EVENTS:
Time Frame: 9 months
Description: All adverse events experienced by participants were collected from the time of the first dose of study treatment, through the study and until the final study visit.
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=6)
delirium (Psychiatric disorders) | 1
myocarditis (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=6)
sinus tachycardia (Cardiac disorders) | 3
diarrhea (Gastrointestinal disorders) | 6
mucositis - oral (Gastrointestinal disorders) | 4
nausea (Gastrointestinal disorders) | 6
vomiting (Gastrointestinal disorders) | 5
fatigue (General disorders) | 6
elevated alanine aminotransferase (Investigations) | 3
elevated aspartate aminotransferase (Investigations) | 3
blood bilirubin increased (Investigations) | 2
arthralgia (Musculoskeletal and connective tissue disorders) | 6
myalgia (Musculoskeletal and connective tissue disorders) | 3
cognitive disturbance (Nervous system disorders) | 1
headache (Nervous system disorders) | 2
delirium (Psychiatric disorders) | 2
erythroderma (Skin and subcutaneous tissue disorders) | 2
rash acneiform (Skin and subcutaneous tissue disorders) | 3
rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
capillary leak syndrome (Vascular disorders) | 3
hypotension (Vascular disorders) | 4
acute kidney injury (Renal and urinary disorders) | 2
acidosis (Renal and urinary disorders) | 4
Platelet count decreased (Investigations) | 1
Infection - C. difficile (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
The protocol terminated early due to a dramatic change in the treatment landscape for treating BRAF mutant melanoma (e.g. one BRAF/MEK inhibitor combination and two anti-PD1 antibodies were approved by the FDA while this study was open).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes